CLINICAL TRIAL: NCT06453070
Title: Hasan Kalyoncu University
Acronym: HKU
Status: Completed | Type: Observational
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Eda Atay, Research Assitant, Hasan Kalyoncu University
Other Study IDs: HKUU; Fırat University (Other: Fırat University)
Record Dates: First submitted 2024-06-07; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Aggression; Forensic Psychiatric Patients
Keywords: Forensic Psychiatric Patients; Aggression; childhood traumas; cognitive distortions; nursing
MeSH Terms: conditions — Aggression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention was made — No intervention was made

SUMMARY:
Aggression is a serious problem that appears to be common in forensic psychiatric patients. Determining factors related to aggression is important for psychiatric nurses during the treatment, care and rehabilitation of patients. The aim of this study is to determine the relationship between childhood traumas, cognitive distortions and aggression in forensic psychiatry patients. This descriptive study was conducted with 103 male forensic psychiatry patients treated in a high security forensic psychiatry hospital. The data of study were collected Introductory Information Form, Childhood Psychological Traumas Scale (CTQ), Cognitive Distortions Scale (CDS) and Buss-Perry Aggression Scale (BAQ). In this study, 82.5% of forensic psychiatry patients were male, 50.5% were married, 49.5% had secondary education, 53.4% were not working. It was found that patients diagnosed with Schizophrenia Spectrum and Other Psychotic Disordersa and Bipolar Affective Disorders, who were hospitalised more than 5 times, who used alcohol/substances and who had previous experience of forensic events had higher levels of aggression. There was a significant positive correlation between the childhood traumas, cognitive distortions and aggression. The results of this study reveal important results that will contribute to psychiatric nurses caring for forensic psychiatric patients in determining the patients' aggression and affecting factors during the treatment and care process.

ELIGIBILITY:
Inclusion Criteria:

* people who do not have criminal liability
* do not have a reading comprehension problem
* volunteers to participate in the research

Exclusion Criteria:

* Patients who did not agree to participate in the study or who left the study

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: They are people who do not have criminal liability, do not have a reading comprehension problem, and volunteer to participate in the research. Since the forensic women's service was not active, the sample consisted of 103 male patients.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
There was a significant correlation between the childhood traumas and aggression | Four mounth
There was a significant correlation between the cognitive distortions and aggression | Four mounth

CONTACTS AND LOCATIONS:
Locations (1):
- Forensic Psychiatry Unit of Elazığ Fethi Sekin City Hospital, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No